CLINICAL TRIAL: NCT02836002
Title: 'Controlled Human Malaria Infection Study to Assess Gametocytaemia and Mosquito Transmissibility in Participants Challenged With Plasmodium Falciparum by Sporozoite Challenge to Establish a Model for the Evaluation of Transmission-blocking Interventions'
Brief Title: Controlled Human Malaria Infection Model for Evaluation of Transmission-Blocking Interventions - Study 1
Acronym: CHMI-trans1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); QIMR Berghofer Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHMI-trans1
Record Dates: First submitted 2016-07-06; First posted 2016-07-18 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2017-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; piperaquine; atovaquone, proguanil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 - SP low/SP high (Experimental): Group 1 will be treated with a course of subcurative sulfadoxine-pyrimethamine (SP) (SP low, 500mg/25mg) as treatment 1.
  As treatment 2 (SP high) volunteers will receive a treatment with sulfadoxine-pyrimethamine (1000mg/50mg).
  Group 1 will receive a malaria challenge infection, P. falciparum 3D7 -infected mosquito bites Final treatment with a curative regimen of atovaquone/proguanil (malarone).
  Interventions: Drug: Sulfadoxine-pyrimethamine (low dose); Drug: Sulfadoxine-pyrimethamine (high dose); Biological: malaria challenge infection, P. falciparum 3D7; Drug: Atovaquone-proguanil
- Group 2 - SP low/Pip high (Experimental): Group 2 will be treated with a course of subcurative sulfadoxine-pyrimethamine (SP) (SP low, 500mg/25mg) as treatment 1.
  As treatment 2 (Pip high) volunteers will receive a treatment with piperaquine (960mg).
  Group 2 will receive a malaria challenge infection, P. falciparum 3D7 -infected mosquito bites Final treatment with a curative regimen of atovaquone/proguanil (malarone).
  Interventions: Drug: Sulfadoxine-pyrimethamine (low dose); Drug: Piperaquine (high dose); Biological: malaria challenge infection, P. falciparum 3D7; Drug: Atovaquone-proguanil
- Group 3 - Pip low/Pip high (Experimental): Group 3 will receive piperaquine (Pip) in a low-dose (Pip low, 480 mg) as treatment 1.
  As treatment 2 (Pip high) volunteers will receive a treatment with piperaquine (960mg).
  Group 3 will receive a malaria challenge infection, P. falciparum 3D7 -infected mosquito bites Final treatment with a curative regimen of atovaquone/proguanil (malarone).
  Interventions: Drug: Piperaquine (low dose); Drug: Piperaquine (high dose); Biological: malaria challenge infection, P. falciparum 3D7; Drug: Atovaquone-proguanil
- Group 4 - Pip low/SP high (Experimental): Group 4 will receive piperaquine (Pip) in a low-dose (Pip low, 480 mg) as treatment 1.
  As treatment 2 (SP high) volunteers will receive a treatment with sulfadoxine-pyrimethamine (1000mg/50mg).
  Group 4 will receive a malaria challenge infection, P. falciparum 3D7 -infected mosquito bites Final treatment with a curative regimen of atovaquone/proguanil (malarone).
  Interventions: Drug: Piperaquine (low dose); Drug: Sulfadoxine-pyrimethamine (high dose); Biological: malaria challenge infection, P. falciparum 3D7; Drug: Atovaquone-proguanil

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine (low dose) — - subcurative regimen (500mg/25mg)
  Other Names: Fansidar
  Arms: Group 1 - SP low/SP high; Group 2 - SP low/Pip high
Drug: Piperaquine (low dose) — - subcurative regimen (480 mg)
  Other Names: piperaquine phosphate
  Arms: Group 3 - Pip low/Pip high; Group 4 - Pip low/SP high
Drug: Sulfadoxine-pyrimethamine (high dose) — - curative regimen (1000mg/50mg)
  Other Names: Fansidar
  Arms: Group 1 - SP low/SP high; Group 4 - Pip low/SP high
Drug: Piperaquine (high dose) — - curative regimen (960 mg)
  Other Names: piperaquine phosphate
  Arms: Group 2 - SP low/Pip high; Group 3 - Pip low/Pip high
Biological: malaria challenge infection, P. falciparum 3D7 — malaria challenge infection by P. falciparum 3D7-infected mosquito bites
  Other Names: 3D7 Plasmodium falciparum
Drug: Atovaquone-proguanil — - curative regimen: 1000/400 mg, for 3 days
  Other Names: Malarone

SUMMARY:
This is a single-center, open label study. The primary aim of this project is to develop a controlled human malaria infection transmission model ("CHMI-trans") or "challenge model" to evaluate the capacity of vaccines, biologics (monoclonal antibodies, or mAbs), and drugs to block malaria parasite transmission by assessing infectiousness of Plasmodium falciparum (Pf) gametocyte carriers for Anopheles mosquitoes.

DETAILED DESCRIPTION:
A total of 32 volunteers will be randomly assigned to four groups (n=8) and subjected to a standard controlled human malaria infection (CHMI) delivered by five Pf-infected mosquitoes (3D7 clone). Treatment is subsequently initiated to induce gametocytaemia (treatment 1, DT1) and to clear pathogenic asexual parasites whilst leaving gametocytes unaffected (treatment 2, DT2). At the end of the study, treatment of all parasite stages is provided following national treatment guidelines (end treatment, ET).

Once malaria infections are detected by 18S qPCR positive (day of treatment 1 [DT1]), groups 1 and 2 will be treated with a course of subcurative sulfadoxine-pyrimethamine (SP) (SP low, 500mg/25mg). Groups 3 and 4 will receive piperaquine (Pip) in a low-dose (Pip low, 480 mg). After DT1, volunteers will receive a curative treatment (DT2) when a recrudescence of asexual parasitaemia occurs or on day 21 post challenge infection, whichever comes first. Volunteers in group 1 (SP low/SP high) will be treated with sulfadoxine-pyrimethamine (1000mg/50mg) and group 2 (SP low/Pip high) with piperaquine (960mg). Volunteers in group 3 (Pip low/Pip high) will be treated with piperaquine (960mg) and group 4 (Pip low/SP high) with sulfadoxine-pyrimethamine (1000mg/50mg). To ensure the radical clearance of all parasite stages, all volunteers will receive a final treatment (ET) according to national guidelines with atovaquone/proguanil (Malarone®) on day 42. Daily blood samples will allow detailed quantification of gametocytes, gametocyte sex ratio and ex vivo assessments of gametocyte fitness.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Subject is aged ≥ 18 and ≤ 35 years and in good health.
2. Subject has adequate understanding of the procedures of the study and is able and willing (in the investigator's opinion) to comply with all study requirements.
3. Subject is willing to complete an informed consent questionnaire and is able to answer all questions correctly.
4. Subject is able to communicate well with the investigator and is available to attend all study visits, lives in proximity to the trial centre (<10 km) or (if >10km) is willing to stay in a hotel close to the trial centre during part of the study (from day 5 post-infection until DT1+4 provided that the subject has had 2 consecutive negative 18S qPCR tests (at least 24 hours apart) following DT1 treatment; or until day DT2+3).
5. The subject will remain within the Netherlands during the challenge period, will not travel to a malaria-endemic area during the study period, and is reachable (24/7) by mobile telephone throughout the entire study period.
6. Subject agrees to their general practitioner being informed and contacted about their participation in the study and agrees to sign a form to request the release by their General Practitioner (GP), and medical specialist when necessary, to the investigator(s), of any relevant medical information concerning possible contra-indications for participation in the study.
7. The subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period and for a defined period thereafter according to current Sanquin guidelines.
8. For female subjects: subject agrees to use continuous adequate contraception** and not to breastfeed for the duration of study.
9. Subject agrees to refrain from intensive physical exercise (disproportionate to the subjects usual daily activity or exercise routine) during the malaria challenge period.
10. Subject has signed written informed consent to participate in the trial.

(*Acceptable forms of contraception include: established use of oral, injected or implanted hormonal contraceptives; intrauterine device or intrauterine system; barrier methods (condoms or diaphragm with additional spermicide); male partner's sterilisation (with appropriate post-vasectomy documentation of absence of sperm in the ejaculate); true abstinence when this is in line with the preferred and usual lifestyle of the subject; Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following.

   1.1. Body weight <50 kg or Body Mass Index (BMI) <18 or >30 kg/m2 at screening. 1.2. A heightened risk of cardiovascular disease, as determined by: an estimated ten year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.

   1.3. A medical history of functional asplenia, sickle cell trait/disease, thalassaemia trait/disease or G6PD-deficiency.

   1.4. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   1.5. Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) 1.6. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.

   1.7. Any recent or current systemic therapy with an antibiotic or drug with potential anti-malarial activity (chloroquine, doxycycline, tetracycline, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, erythromycin, hydroxychloroquine, etc.) (allowable timeframe for use at the Investigator's discretion).

   1.8. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.

   1.9. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

   1.10. History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or at inclusion, or positive urine toxicology test for cannabis at inclusion.
2. For female subjects: positive urine pregnancy test at screening and/or at the baseline visit.
3. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study.
4. Known hypersensitivity to or contra-indications (including co-medication) for use of sulfadoxine-pyrimethamine, piperaquine, chloroquine, Malarone®, artemether-lumefantrine, primaquine or history of severe (allergic) reactions to mosquito bites.
5. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
6. Being an employee or student of the department of Medical Microbiology of the Radboudumc or the department of Internal Medicine.
7. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Frequency and magnitude of adverse events in the CHMI-trans model in study groups | up to day 42 after challenge infection
  Frequency and magnitude of adverse events in the CHMI-trans model in study groups.
gametocyte prevalence | up to day 42 after challenge infection
  Prevalence of gametocytes in the CHMI-trans model in study groups.

SECONDARY OUTCOMES:
peak density gametocytes | up to day 42 after challenge infection
  Peak density and time-point of peak density of gametocytes by qRT-PCR.
AUC gametocytes | up to day 42 after challenge infection
  The area under the curve of gametocyte density versus time.
Gametocyte sex-ratio | up to day 42 after challenge infection
  ratio of male-female gametes

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] Reuling IJ, van de Schans LA, Coffeng LE, Lanke K, Meerstein-Kessel L, Graumans W, van Gemert GJ, Teelen K, Siebelink-Stoter R, van de Vegte-Bolmer M, de Mast Q, van der Ven AJ, Ivinson K, Hermsen CC, de Vlas S, Bradley J, Collins KA, Ockenhouse CF, McCarthy J, Sauerwein RW, Bousema T. A randomized feasibility trial comparing four antimalarial drug regimens to induce Plasmodium falciparum gametocytemia in the controlled human malaria infection model. Elife. 2018 Feb 27;7:e31549. doi: 10.7554/eLife.31549. PMID 29482720
- [Derived] Post A, Kabore B, Reuling IJ, Bognini J, van der Heijden W, Diallo S, Lompo P, Kam B, Herssens N, Lanke K, Bousema T, Sauerwein RW, Tinto H, Jacobs J, de Mast Q, van der Ven AJ. The XN-30 hematology analyzer for rapid sensitive detection of malaria: a diagnostic accuracy study. BMC Med. 2019 May 31;17(1):103. doi: 10.1186/s12916-019-1334-5. PMID 31146732
- Available data/document: Individual Participant Data Set — https://datadryad.org//resource/doi:10.5061/dryad.60h41